CLINICAL TRIAL: NCT07407985
Title: A Open-label, Single-arm Clinical Trial Designed to Evaluate the Safety, Pharmacokinetic , and Efficacy of the GK01 Cell Injection in Combination With a PD-1 Monoclonal Antibody for the Treatment of Advanced Solid Tumors.
Brief Title: A Clinical Study to Evaluate GK01 Cell Injection in Combination With PD-1 Monoclonal Antibody for Advanced Solid Tumors
Acronym: GK01IIT-TZ03
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Beijing Geekgene Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUARDIAN-03
Record Dates: First submitted 2026-01-11; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GK01 PD-1 monoclonal (Experimental): GK01 combination with PD-1 monoclonal antibody
  Interventions: Drug: GK01 combination with PD-1 monoclonal antibody

INTERVENTIONS:
Drug: GK01 combination with PD-1 monoclonal antibody — GK01 combination with PD-1 monoclonal antibody

SUMMARY:
This study is a open-label, single-arm clinical trial designed to evaluate the safety, pharmacokinetic profile, and preliminary efficacy of the GK01 cell injection in combination with a PD-1 monoclonal antibody for the treatment of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) .
* Aged 18 to 70 years (inclusive) at the time of signing the ICF.
* Histologically or cytologically confirmed advanced solid tumors that are metastatic or locally recurrent (including but not limited to small cell lung cancer, non-small cell lung cancer, gastric cancer, colorectal cancer, etc.);
* ECOG score of 0 ~1 .
* Expected survival time is more than 12 weeks.
* Negative blood pregnancy test for females of childbearing potential is required.

Exclusion Criteria:

* Patients with central nervous system (CNS) metastasis, leptomeningeal disease, or metastatic spinal cord compression; or a history of CNS disorders, including but not limited to epilepsy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, etc.
* History of bone marrow or organ transplantation;
* History of other primary malignancies within 5 years prior to study treatment
* Hepatitis B surface antigen (HBsAg) positivity; With negative HBsAg but positive hepatitis B core antibody (HBcAb) ,and if peripheral blood hepatitis B virus (HBV) DNA positive; Hepatitis C virus (HCV) antibody positive and HCV RNA positive; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive; Both Treponema pallidum-specific and non-specific antibody tests are positive.
* Patients with a known allergy to any component of the study drugs.
* Received treatment with anti-PD-1, anti-PD-L1 therapeutic antibodies, or drugs targeting this pathway.
* Received any investigational drug or systemic anticancer therapy within 28 days before infusion (or 5 half-lives of the drug, whichever is considered more appropriate by the investigator).
* Received wide-field radiotherapy within 28 days prior to signing the ICF, with the exception of palliative radiotherapy to non-target lesions for symptom relief, administered at least 14 days before signing the ICF or planned during the study period.
* Undergone major surgery within 28 days prior to signing the ICF, or are scheduled to undergo major surgery during the study period.
* At the time of signing the ICF, any toxicity from prior anti-cancer therapy (except alopecia and pigmentation) that has not recovered to Grade 1 (excluding lymphocytopenia) or to baseline level (according to NCI CTCAE version 5.0).
* Any uncontrolled active infection requiring parenteral (IV) antibiotic, antiviral, or antifungal treatment at the time of signing the ICF or within 4 weeks before the first infusion.
* History of active tuberculosis infection within 1 year prior to screening (subjects with a history of active tuberculosis infection more than 1 year ago are eligible if, in the investigator's judgment, there is no current evidence of active tuberculosis).
* Concurrent or previous history of interstitial lung disease or interstitial pneumonia; presence of chronic lung disease or other respiratory conditions that significantly impair lung function.
* Diagnosis of active autoimmune disease or a history of autoimmune disease that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, psoriasis, etc.), or at risk of such conditions.
* Required treatment with systemic corticosteroids (at a dose equivalent to or higher than 10 mg/day of prednisone) or other immunosuppressive medications within 2 weeks before signing the ICF or during the study period.
* Clinically significant thyroid dysfunction as assessed by the investigator.
* Clinically significant cardiovascular diseases.
* Insufficient bone marrow reserve or insufficient organ function.
* Bleeding within 6 months before signing the ICF; clinically significant bleeding requiring medical intervention within 28 days before screening, including esophageal variceal bleeding.
* Poorly controlled pleural, peritoneal, or pericardial effusion during the screening period (e.g., presence of clinical symptoms, fluctuating volume, requiring repeated drainage, or the use of oral diuretics). Presence of ascites detectable on physical examination, clinical symptoms caused by ascites, or the need for special management such as repeated drainage or intraperitoneal drug infusion (subjects with only a small amount of ascites detectable solely via imaging may be considered for enrollment).
* Administration of attenuated or inactivated vaccines within 28 days before signing the ICF, or planned administration of such vaccines during the screening period.
* The investigator considers that the subject's complications or other conditions may affect compliance with the protocol or that the subject is unsuitable for participation in this study.
* Female subjects who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-12-03 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 years
  The incidence and severity of AEs (Adverse Events) and SAEs (Serious Adverse Events).

SECONDARY OUTCOMES:
Pharmacokinetic | 2 years
  Levels of T-cell Receptor copies
Objective response rate (ORR) | 2 years
  Proportion of subjects achieving complete response (CR) and partial response (PR)
Progression-free Survival（PFS） | 2 years
  Time from GK01 treatment to disease progression or death
Duration of Response（DOR） | 2 years
  Time from first documented evidence of confirmed CR or PR until the first documented evidence of disease progression or death, whichever occurs earlier
Overall survival（OS） | 2 years
  Time from GK01 treatment to death
Disease Control Rate（DCR） | 2 years
  Proportion of subjects achieving best response of CR, PR, or SD treated with GK01

OTHER OUTCOMES:
Biomarker | 2 years
  Concentration levels of serum cytokines, tumor markers and other related markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No